CLINICAL TRIAL: NCT05464355
Title: Feasibility Study of the Use of Biomarkers to Detect Perioperative Brain Injury: the Association Between Serum Neurofilament Light Chains, Tau Proteins, Continuous Intra-operative Electroencephalography, and the Development of Post Operative Cognitive Dysfunction After Surgery
Brief Title: Biomarkers Associated With Postoperative Cognitive Dysfunction
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PID16101; 302168 (Other: Integrated Research Application System); Protocol version 13/06/2022 (Other: University of Oxford)
Record Dates: First submitted 2022-07-11; First posted 2022-07-19 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Delirium; Postoperative Cognitive Dysfunction; Cognitive Decline; Cognitive Impairment
Keywords: Electroencephalography; Delirium; Neurofilament light chain; Tau protein
MeSH Terms: conditions — Delirium; Postoperative Cognitive Complications; Cognitive Dysfunction; Charcot-Marie-Tooth disease, Type 1F; Frontotemporal Dementia | interventions — tau Proteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood tests will be disposed of after analysis according to standard laboratory operating procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biomarker monitoring
  Interventions: Procedure: Intraoperative electroencephalography recording; Procedure: Neurofilament light chain measurement; Procedure: Tau protein measurement

INTERVENTIONS:
Procedure: Intraoperative electroencephalography recording — Intraoperative electroencephalography measurements, a non-invasive routine monitoring device used during anaesthesia to measure the brain's electrical activity
  Other Names: EEG recording
Procedure: Neurofilament light chain measurement — Measurement of the level of neurofilament light chain in a blood sample
  Other Names: NfL
Procedure: Tau protein measurement — Measurement of the level of tau protein in a blood sample

SUMMARY:
Loss of cognitive function after major surgery is a significant risk in older people. It can occur acutely in the days after surgery as delirium or in months to years later as a persistent reduction in brain function termed neurocognitive decline. Together these conditions are called post operative cognitive dysfunction (POCD). They can be acutely distressing for patients and are associated with other problems after surgery.

The causes of post operative cognitive dysfunction are poorly understood. Studies have been limited by a lack of biomarkers to predict which patients are at high risk of developing POCD. Research suggests silent strokes occurring during surgery and different sensitivities to anaesthetic medicines are associated with POCD.

The project consists of a feasibility study to investigate markers that might predict people over 65 years old getting POCD. The first biomarker is a non-invasive monitor of anaesthetics effects on brain function called electroencephalography (EEG): The investigators will identify which EEG patterns predict delirium within five days surgery. The second set of biomarkers are two blood tests of proteins that increase after strokes: these are neurofilament light chains and tau proteins. The investigators will establish if these can be used to predict having POCD up to one year after surgery and long term cognitive impairment up to 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 65 years of age
* Having elective non-cardiac surgery under general anaesthesia
* Anticipated to have at least 48 hours of inpatient admission
* Able & willing to give informed consent

Exclusion Criteria:

* Unable to participate in neurocognitive assessments
* Presence of delirium prior to surgery
* Contraindication to use of EEG electrodes (e.g. known allergy to a component of the electrodes)
* Known history of severe traumatic brain injury
* Learning disability specifically with a known structural brain lesion
* Known history of dementia
* Participants undergoing operations on the carotid artery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults over 65 years of age having major elective surgery under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility to conduct the study | 1 year after surgery
  The total number of participants who are successfully recruited, receive the study procedures and complete both 90 day and 1 year follow up after surgery.

SECONDARY OUTCOMES:
Postoperative delirium incidence and severity | Up to 5 days after surgery
  Postoperative delirium identified as being present according to a positive result using 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) and severity according to the absolute value on the 3D-CAM-Severity which is a scale converting the 3-Minute Diagnostic Interview for Confusion Assessment Method into a scale from 0-7. Higher scores are associated with worse outcome.
Days alive and at home up to 90 days after surgery | 90 days after surgery
  The number of days a participant is alive and how many are spent at home after surgery
Change in neurofilament light chains and tau proteins levels pre- to post operatively | Up to 2 days after surgery
  Measurements of the level of the biomarkers neurofilament light chain and tau protein in plasma
Postoperative neurocognitive dysfunction and severity | Up to 1 year after surgery
  Cognitive impairment measured on Montreal Objective Cognitive Assessment administered by telephone. The scale is 0-22 with higher scores representing better outcome.
Long term cognitive impairment | Up to 5 years after surgery
  Incidence of new diagnosis in primary or secondary care of dementia or mild cognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: Martyn Ezra, Principal Investigator — University of Oxford
Locations (1):
- Royal Berkshire NHS Foundation Trust, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Participants will be asked for consent to share anonymized data with other researchers.